CLINICAL TRIAL: NCT00196560
Title: A Randomized Evaluation of Immobilization in External Rotation in the Management of Acute Anterior Dislocations of the Shoulder
Brief Title: Immobilization in External Rotation of Acute Shoulder Dislocations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fowler Kennedy Sport Medicine Clinic (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); American Shoulder and Elbow Surgeons (Other)
Responsible Party: Principal Investigator, Sharon Griffin, Research Coordinator, Fowler Kennedy Sport Medicine Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKSMC PSI ERAADS
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Anterior Shoulder Dislocation
Keywords: Immobilization in External Rotation; Acute primary anterior shoulder dislocation
MeSH Terms: interventions — Immobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- exernal rotation (Experimental): external rotation at 90 degrees
  Interventions: Device: Immobilization in External Rotation

INTERVENTIONS:
Device: Immobilization in External Rotation

SUMMARY:
The purpose of this study is to determine whether immobilizing the affected shoulder of first time anterior shoulder dislocation patients in external rotation (vs immobilization in traditional internal rotation) reduces the rate of recurrent dislocations experienced in 24 months.

DETAILED DESCRIPTION:
Immobilizing the affected shoulder of first time anterior shoulder dislocation patients in external rotation (vs immobilization in traditional internal rotation)should reduce the rate of recurrent dislocations experienced in 24 months.

ELIGIBILITY:
Inclusion Criteria:

* skeletally mature patients less than 30 years of age
* sustained an acute, first-time, traumatic anterior dislocation of the shoulder as defined by; i. Mechanism of abduction, external rotation ii. Sudden pain in the shoulder iii. Manipulative reduction required or iv. Radiograph documenting a dislocated joint
* willing to participate in follow-up for at least two years

Exclusion Criteria:

* incompetent or unwilling to consent
* inability or unwillingness to comply with rehabilitative protocol or required follow-up assessments
* previous instability of the affected shoulder
* significant associated fracture (exception Hill Sachs or Bankart lesions)
* concomitant ipsilateral upper extremity injuries which may affect the patient's ability to participate in, or benefit from, a rehabilitative program
* a history of significant ligamentous laxity or demonstrated multi-directional instability of the contralateral shoulder
* neurovascular compromise of the affected limb
* a medical condition making the patient unable to wear a brace or sling

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2003-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Recurrent Instability at 24 months

SECONDARY OUTCOMES:
Time (weeks) to return to work and time(weeks) to return to sport
Complications (resulting from immobilization)
Compliance with immobilization protocol
Western Ontario Shoulder Instability index (WOSI)
American Shoulder and Elbow Surgeons questionnaire (ASES)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Litchfield, MD, FRCS(C), Principal Investigator — Fowler Kennedy Sport Medicine Clinic
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, London, Ontario, Canada

REFERENCES:
- [Background] Kazar B, Relovszky E. Prognosis of primary dislocation of the shoulder. Acta Orthop Scand. 1969;40(2):216-24. doi: 10.3109/17453676908989501. No abstract available. PMID 5365161
- [Background] ROWE CR. Prognosis in dislocations of the shoulder. J Bone Joint Surg Am. 1956 Oct;38-A(5):957-77. No abstract available. PMID 13367074
- [Background] Kirkley A, Griffin S, McLintock H, Ng L. The development and evaluation of a disease-specific quality of life measurement tool for shoulder instability. The Western Ontario Shoulder Instability Index (WOSI). Am J Sports Med. 1998 Nov-Dec;26(6):764-72. doi: 10.1177/03635465980260060501. PMID 9850776
- [Background] Aronen JG, Regan K. Decreasing the incidence of recurrence of first time anterior shoulder dislocations with rehabilitation. Am J Sports Med. 1984 Jul-Aug;12(4):283-91. doi: 10.1177/036354658401200408. PMID 6476187
- [Background] Henry JH, Genung JA. Natural history of glenohumeral dislocation--revisited. Am J Sports Med. 1982 May-Jun;10(3):135-7. doi: 10.1177/036354658201000301. PMID 7114346
- [Background] Bottoni CR, Wilckens JH, DeBerardino TM, D'Alleyrand JC, Rooney RC, Harpstrite JK, Arciero RA. A prospective, randomized evaluation of arthroscopic stabilization versus nonoperative treatment in patients with acute, traumatic, first-time shoulder dislocations. Am J Sports Med. 2002 Jul-Aug;30(4):576-80. doi: 10.1177/03635465020300041801. PMID 12130413
- [Background] Rowe CR, Patel D, Southmayd WW. The Bankart procedure: a long-term end-result study. J Bone Joint Surg Am. 1978 Jan;60(1):1-16. PMID 624747
- [Background] Hovelius L, Augustini BG, Fredin H, Johansson O, Norlin R, Thorling J. Primary anterior dislocation of the shoulder in young patients. A ten-year prospective study. J Bone Joint Surg Am. 1996 Nov;78(11):1677-84. doi: 10.2106/00004623-199611000-00006. PMID 8934481
- [Background] McLaughlin HL, MacLellan DI. Recurrent anterior dislocation of the shoulder. II. A comparative study. J Trauma. 1967 Mar;7(2):191-201. doi: 10.1097/00005373-196703000-00002. No abstract available. PMID 6018942
- [Background] Simonet WT, Cofield RH. Prognosis in anterior shoulder dislocation. Am J Sports Med. 1984 Jan-Feb;12(1):19-24. doi: 10.1177/036354658401200103. PMID 6703178
- [Background] Wheeler JH, Ryan JB, Arciero RA, Molinari RN. Arthroscopic versus nonoperative treatment of acute shoulder dislocations in young athletes. Arthroscopy. 1989;5(3):213-7. doi: 10.1016/0749-8063(89)90174-6. PMID 2775396
- [Background] DeBerardino TM, Arciero RA, Taylor DC, Uhorchak JM. Prospective evaluation of arthroscopic stabilization of acute, initial anterior shoulder dislocations in young athletes. Two- to five-year follow-up. Am J Sports Med. 2001 Sep-Oct;29(5):586-92. doi: 10.1177/03635465010290051101. PMID 11573917
- [Background] Arciero RA, Wheeler JH, Ryan JB, McBride JT. Arthroscopic Bankart repair versus nonoperative treatment for acute, initial anterior shoulder dislocations. Am J Sports Med. 1994 Sep-Oct;22(5):589-94. doi: 10.1177/036354659402200504. PMID 7810780
- [Background] Kirkley A, Griffin S, Richards C, Miniaci A, Mohtadi N. Prospective randomized clinical trial comparing the effectiveness of immediate arthroscopic stabilization versus immobilization and rehabilitation in first traumatic anterior dislocations of the shoulder. Arthroscopy. 1999 Jul-Aug;15(5):507-14. doi: 10.1053/ar.1999.v15.015050. PMID 10424554
- [Background] Arciero RA. Acute arthroscopic Bankart repair? Knee Surg Sports Traumatol Arthrosc. 2000;8(2):127-9. doi: 10.1007/s001670050199. No abstract available. PMID 10795677
- [Background] Eriksson E. Should first-time traumatic shoulder dislocations undergo an acute stabilization procedure? Knee Surg Sports Traumatol Arthrosc. 2003 Mar;11(2):61-2. doi: 10.1007/s00167-003-0357-8. No abstract available. PMID 12884846
- [Background] Kirkley A, Werstine R, Ratjek A, Griffin S. Prospective randomized clinical trial comparing the effectiveness of immediate arthroscopic stabilization versus immobilization and rehabilitation in first traumatic anterior dislocations of the shoulder: long-term evaluation. Arthroscopy. 2005 Jan;21(1):55-63. doi: 10.1016/j.arthro.2004.09.018. PMID 15650667
- [Background] Itoi E, Sashi R, Minagawa H, Shimizu T, Wakabayashi I, Sato K. Position of immobilization after dislocation of the glenohumeral joint. A study with use of magnetic resonance imaging. J Bone Joint Surg Am. 2001 May;83(5):661-7. doi: 10.2106/00004623-200105000-00003. PMID 11379734
- [Background] Itoi E, Hatakeyama Y, Kido T, Sato T, Minagawa H, Wakabayashi I, Kobayashi M. A new method of immobilization after traumatic anterior dislocation of the shoulder: a preliminary study. J Shoulder Elbow Surg. 2003 Sep-Oct;12(5):413-5. doi: 10.1016/s1058-2746(03)00171-x. PMID 14564258
- [Background] Arciero RA, DeBernadino TM. Acute and chronic dislocations of the shoulder. In Norris TR (ed), Orthopaedic Knowledge update: Shoulder and Elbow. Rosemont Il, American Academy of Orthopaedic Surgeons, 1997, pp 69-71.
- [Background] Donner, A. Epidemiology 560B course notes. UWO, January 2003.
- [Background] Michener LA, McClure PW, Sennett BJ. American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form, patient self-report section: reliability, validity, and responsiveness. J Shoulder Elbow Surg. 2002 Nov-Dec;11(6):587-94. doi: 10.1067/mse.2002.127096. PMID 12469084
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738
- [Derived] Whelan DB, Litchfield R, Wambolt E, Dainty KN; Joint Orthopaedic Initiative for National Trials of the Shoulder (JOINTS). External rotation immobilization for primary shoulder dislocation: a randomized controlled trial. Clin Orthop Relat Res. 2014 Aug;472(8):2380-6. doi: 10.1007/s11999-013-3432-6. PMID 24385033